CLINICAL TRIAL: NCT04003688
Title: Strategy to Calculate Magnesium Sulfate Dose in Obese Patients. A Randomized and Blind Trial.
Brief Title: Magnesium Sulfate Dose in Obese Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Joaquim Edson Vieira, Associate professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAAE 09006119.2.0000.5501
Record Dates: First submitted 2019-06-24; First posted 2019-07-01 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Magnesium Sulfate; Postoperative Pain; Obesity
MeSH Terms: conditions — Pain, Postoperative; Obesity

STUDY DESIGN:
Intervention Model Description: Prospective, double-blind, randomized clinical trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The anesthesiologist in charge of randomization will number 75 opaque envelopes and insert a card in each with the corresponding information of the group (according to the lottery) and the medication to be administered. Another anesthesiologist in charge of preparing the blind solution alone will open the envelope. Both of these investigators, as well as the anesthesiologist providing anesthesia and the anesthesiologist in charge of data evaluation will not participate in any of the other steps of the trial. The patients will be blinded to their own treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Patient will be administered saline solution followed by venous general anesthesia.
  Interventions: Drug: Placebo group
- Magnesium sulfate through real weight group (Experimental): Patient will be administered magnesium sulfate 40 mg/kg of the patient's actual weight followed by venous general anesthesia.
  Interventions: Drug: Magnesium sulfate through real weight group
- Magnesium sulfate through ideal corrected weight group (Experimental): Patient will be administered magnesium sulfate 40 mg/kg of the patient's ideal corrected weight followed by venous general anesthesia.
  Interventions: Drug: Magnesium sulfate through ideal corrected weight group

INTERVENTIONS:
Drug: Magnesium sulfate through real weight group — Magnesium sulfate dose 40 mg/kg of actual patient's weight
  Other Names: Real weight group
  Arms: Magnesium sulfate through real weight group
Drug: Placebo group — Saline solution (instead of magnesium sulfate, as in the other groups)
  Arms: Placebo group
Drug: Magnesium sulfate through ideal corrected weight group — Magnesium sulfate dose 40 mg/kg of ideal corrected patient's weight
  Other Names: Ideal weight group
  Arms: Magnesium sulfate through ideal corrected weight group

SUMMARY:
Magnesium sulfate has been applied in various situations due to actual or potential benefits related to neuroprotection, treatment of eclampsia/pre-eclampsia, arterial hypertension, adrenergic reflex under laryngoscopy/intubation and, shivering, nausea and vomiting, among others. In anesthesia it has been useful as an analgesic adjuvant; however, the method to calculate the dose of magnesium sulfate in obese population is unclear. The objective of this project is to compare two methods of dose calculation based either on the real weight or corrected ideal weight.

DETAILED DESCRIPTION:
Magnesium sulfate has been applied in various situations due to actual or potential benefits related to neuroprotection, treatment of eclampsia/pre-eclampsia, arterial hypertension, adrenergic reflex under laryngoscopy/intubation and, shivering, nausea and vomiting, among others. In anesthesia it has been useful as an analgesic adjuvant; however, the method to calculate the dose of magnesium sulfate in obese population is unclear. The objective of this project is to compare two methods of dose calculation based either on the real weight or corrected ideal weight.

Main objective: To determine the optimum strategy to safely and effectively obtain the value of magnesium concentration in the blood of obese population.

Secondary objectives: To evaluate postoperative analgesia and the pharmacokinetic profile of neuromuscular blocker used in each group.

Hypothesis: The null hypothesis is that no matter which method we use to calculate the magnesium sulfate dosage, the blood magnesium concentration will be the same. The alternative hypothesis is that magnesium sulfate dosage based on the patient's actual weight generates higher concentrations of magnesium than that required for postoperative analgesia, as compared with dosage based on that corrected ideal weight of the patient.

Trial design: this is a prospective, controlled, randomized and double-blind clinical trial.

Study setting This study will be conducted at Beneficence Portuguese Society, Santos, an academic hospital, in São Paulo, Brazil. A sample of 75 participants will be recruited from a population of obese patients scheduled to undergo cholecystectomy or bariatric surgery through laparoscopy.

Interventions In the first phase of the trial, 10 patients with body mass index 20-30 kg/m² will be administered magnesium sulphate 40 mg/kg at anesthetic induction. In all patients, blood collection will be conducted before administration of magnesium sulfate, and at 15, 30, 60, 120 and 240 minutes after administration of magnesium sulfate.

In the second phase of the trial, from among obese patients scheduled to undergo cholecystectomy or bariatric surgery through laparoscopy at our institute, 75 patients will be invited to participate in the trial. Participants will be assigned to three groups by electronic randomization process as follow: Placebo group (PG) without administration of magnesium sulfate; real weight group (RWG) administration of magnesium sulfate at 40 mg/kg of the patient's actual weight; corrected ideal weight group (CWG) administration of magnesium sulphate at 40 mg/kg of patient's corrected ideal weight.

The corrected ideal weight will be calculated using the following formulas:

Ideal weight Man = height (cm) - 100 Woman = height (cm) - 105 Corrected ideal weight = Ideal weight + (0,4 x difference between the real and ideal weight) The participants will not be administered any sedative agent before anesthetic induction. At arrival in the operating room, all patients will undergo electrocardiography, noninvasive blood pressure measurement, pulse oximetry, monitoring of neuromuscular function, and that of the level of consciousness. Venous access and hydration will be achieved according to the anesthesiologist's judgment. At the time of puncture of the vein, the first 2-ml blood sample will be collected to establish the basal concentration of magnesium in the blood. Within 10 min after collection of the blood, dosage will be calculated according to the following chart (Figure 1).

In all participants, infusion of treatment solution will be performed by a blinded investigator, and ketoprofen 100 mg, clonidine 2 µg/kg, cefazolin 2 g, dexamethasone 4 mg, ranitidine 50 mg and lidocaine 1,5 mg/kg will be administered simultaneously. At the end of infusion participants will undergo pre-oxygenation with 100% O2 for 3 to 5 min, followed by propofol through target controlled infusion with initial target of 4 µg/ml according to Marsh's pharmacokinetic model, under monitoring for the level of hypnoses. At the time of adequate level of hypnoses, revealed by the hypnoses monitor (SedLine® Brain Function Monitoring) calibration of the monitor of neuromuscular function (train-of-four - TOF) will be performed; subsequently, cisatracurium 0.15 mg/kg will be administered, and target-controlled infusion of remifentanil (Minto's pharmacokinetic model) at initial target concentration of 5 ng/ml will be conducted. Under hypnoses monitoring, 0.03 mg/kg cisatracurium will be administered if TOF ≥ 2 is observed or on surgical demand. Remifentanil infusion will be conducted according to the patient's hemodynamics, such that systolic pressure is maintained within 30% limits from the baseline value, or maximum value of 130 mmHg and minimum value of 90 mmHg are achieved. During the last 20 minutes' period of surgery, cisatracurium will be withheld, when possible. At the end of surgery, at TOF > 2, atropine 20 µg/kg and neostigmine 40 µg/kg will be administered.

Before extubation, the patients in both groups will be administered morphine 0,05 mg/kg and dipyrone 30 mg/kg. Five minutes after extubation and after each 30 minutes' interval, repeat dose of morphine will be administered at pain-score of > 3 (0 to 10) of the patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 to 60 year-old
* body mass index > 30 kg/m²
* American Society of Anesthesiologists score < III.

Exclusion Criteria:

* Allergy to any medications of the trial
* refusal to participate or sign the consent form
* any global diagnosed neuromuscular disorder
* cardiac conduction blockade higher than atrioventricular block II
* use of illicit drugs, use of calcium channel blockers
* creatinine > 2 mg/dl.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2020-11-12 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Magnesium blood concentration at the preset timepoints. | Four hours
  Comparison of the magnesium concentration (mg/ml) in blood between groups

SECONDARY OUTCOMES:
Opioid consumption | Four hours.
  Opioid consumption (microgram)
Time to recovery from neuromuscular blockade | During recovery time (just after the end of surgery)
  Time between cisatracurium administration (last dose) and train-of-four monitoring 90% (in minutes)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquim Vieira, Professor, Principal Investigator — University of Sao Paulo School of Medicine; Sebastião Silva Filho, Physician, Study Chair — University of Sao Paulo School of Medicine
Locations (1):
- Hospital das Clínicas - Faculdade de Medicina da Universidade de Sao Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data.